CLINICAL TRIAL: NCT02249442
Title: An Open-label Study to Determine the Pharmacokinetics of Single-dose and/or Steady-state TPV/r 500/200 mg in Subjects With Mild and Moderate Hepatic Insufficiency
Brief Title: Study to Determine the Pharmacokinetics on TPV/r in Subjects With Mild and Moderate Hepatic Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.32
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — tipranavir; Ritonavir

ARMS (2):
- Scheme A, mild hepatic subjects (Experimental): multi-dose
  Interventions: Drug: Tipranavir (TPV); Drug: Ritonavir (r)
- Scheme B, moderate hepatic subjects (Experimental): single dose
  Interventions: Drug: Tipranavir (TPV); Drug: Ritonavir (r)

INTERVENTIONS:
Drug: Tipranavir (TPV)
Drug: Ritonavir (r)

SUMMARY:
To determine the pharmacokinetics of single-dose and steady-state Tipranavir/Ritonavir (TPV/r) 500/200 mg in subjects with mild to moderate hepatic insufficiency

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation.
2. Male and female subjects with:

   * Diagnostically established hepatic disease with mild hepatic insufficiency (defined as maximum ever Child-Pugh score ≤6) or
   * Diagnostically established hepatic disease with moderate hepatic insufficiency (defined as maximum ever Child-Pugh score ≤9) for less than 5 years. Current Child-Pugh score must be less than 9 or
   * Subjects matched by gender, race, age (±3 years), and weight (±3 kg) and cigarette smoking (matched where possible by +/- .25 pack years) to subjects with mild or moderate hepatic impairment already enrolled in the study.
3. Body Mass Index (BMI) between 18 and 29 kg/m2
4. Subjects ≥18 and ≤75 years old.
5. Ability to swallow multiple large capsules without difficulty.
6. Laboratory values that indicate adequate baseline organ function are required at the time of screening. All subjects (including healthy controls) should have all laboratory values less than or equal to Grade 1, based on the AIDS Clinical Trial Group (ACTG) Grading Scale.The following exceptions will be made only for subjects with mild or moderate hepatic insufficiency:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 x upper limit normal (ULN) (≤ Grade 2)
   * Alkaline Phosphatase <2 x ULN
   * Hemoglobin >10.0 g / dL
   * Platelets >75,000 / μl
7. Willingness to abstain from alcohol starting 2 days prior to administration of study drug up to the end of the study.
8. Willingness to abstain from the following 72 hours prior to pharmacokinetic (PK) sampling: Garlic supplements, methylxanthine containing drinks (coffee, tea, cola, energy drinks, chocolate, etc.).
9. Willingness to abstain from over the counter herbal medications for the duration of the study.
10. Acceptable medical history, physical examination and chest X-ray (at investigator's discretion) are required prior to entering the treatment phase of the study.
11. Willingness to abstain from the following starting 14 days prior to administration of study drug up until the end of the study: Grapefruit or grapefruit juice; Red wine; Seville oranges (marmalade); St. John's Wort or Milk Thistle.
12. Willingness to abstain from vigorous physical exercise during intense PK study days (Days 1 and 7).
13. Reasonable probability for completion of the study, including dosing requirements of TPV/r and risk for hepatic decompensation among subjects with mild and moderate hepatic insufficiency.

Exclusion Criteria:

1. Female subjects who are of reproductive potential who:

   * Have positive serum β-hCG (Human chorionic gonadotropin test for pregnancy) at Visit 1 or on Day 0.
   * Have not been using a barrier contraceptive method for at least 3 months prior to Day 0 (Visit 2).
   * Are not willing to use a reliable method of at least barrier contraception, during the trial and 60 days after completion/termination.
   * Are breast-feeding.
2. Participation in another trial with an investigational medicine within 60 days prior to Day 0 (Visit 2).
3. Use of any medication listed in the protocol within 30 days prior to Day 0 (Visit 2).
4. Use of any pharmacological contraceptive (including oral or patch) for one month prior to study initiation and for the duration of the study. Use of implantable or injectable contraceptive agents is excluded for at least six months prior to study start.
5. Use of hormone replacement therapy with estrogen-based preparations for at least 1 month prior to study initiation and for the duration of the study.
6. Administration of antimicrobial agents within 10 days prior to Day 0 (Visit 2) or during the trial.
7. Subjects with a history of spontaneous bacterial peritonitis, advanced hepatic cirrhosis (including Child's-Pugh score >8), active esophageal variceal disease, or asterixis.
8. Subjects with active or untreated hepatocellular carcinoma or who test positive for serum alpha fetoprotein (>10mg/dL).
9. Subjects with active coagulopathy.
10. Have serological evidence of exposure to, or infection with, HIV.
11. Recent history of alcohol or substance abuse (within 6 months of study period).
12. Blood or plasma donations within 30 days prior to Day 0 (Visit 2).
13. Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min. For subjects with a resting heart rate below 50, or above 90, the investigator could discuss exclusion with the medical monitor on a case-by-case basis.
14. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV and ritonavir (RTV).
15. Subjects who have had an acute illness within 2 weeks prior to Day 0 (Visit 2).
16. Current use of any medications to control symptoms of hepatic disease within 30 days prior to Day 0, (Visit 2) or for the duration of the trial.
17. Known hypersensitivity to TPV, Ritonavir or the sulphonamide class of drugs.
18. Inability to adhere to the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2004-06-01 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of drug in plasma over the time interval from 0 extrapolated to infinity) | Up to day 12 after first drug administration
AUC0-12h (area under the concentration time curve of drug in plasma over the time interval from 0 to 12h) | Up to 12 hours after drug administration
Cmax (maximum concentration of drug in plasma) | Up to day 12 after first drug administration
Cp12h (drug concentration in plasma at 12 hours after administration) for the mild hepatic subjects | Up to 12 hours (h) after drug administration

SECONDARY OUTCOMES:
time from dosing to the maximum concentration (tmax) | Up to day 12 after first drug administration
elimination half-life (t1/2) | Up to day 12 after first drug administration
oral clearance (CL/F) | Up to day 12 after first drug administration
volume of distribution (Vz/F) | Up to day 12 after first drug administration
Relationship between pharmacokinetic parameters and baseline covariates | Up to day 12 after first drug administration
  Covariates = age, weight, race, cigarette smoking and hepatic impairment
Relationship between pharmacokinetic parameters and baseline covariates | Up to day 12 after first drug administration
  Covariates = age, weight, race, cigarette smoking and the child-Pugh score as linear and quadratic terms
Number of patients with abnormal changes in clinical laboratory parameters | Up to day 12 after first drug administration
Number of patients with adverse events | Up to day 12 after first drug administration

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com